CLINICAL TRIAL: NCT03207139
Title: Ga-68 PSMA Ligand: A Radiopharmaceutical for Localization of Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jing-Ren Tseng, Nuclear Medicine, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201600097A0
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Latent Cancer Prostate
Keywords: cancer prostate; Ga-68 PSMA Ligand; staging; biochemical failure
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ga-68 PSMA ligand (Experimental): Diagnostic performance of [Ga68] PSMA-11
  Interventions: Drug: Ga-68 PSMA ligand

INTERVENTIONS:
Drug: Ga-68 PSMA ligand — For PET/CT PSMA ligand scan, the subject will have catheter(s) placed for intravenous administration of [68Ga]PSMA ligand . Subjects will receive a single intravenous bolus of 2-5 mCi [68Ga]PSMA ligand and received PET/CT scan 60 minutes later. The data acquisition begin with non-contrast CT at 120kVp, automated mAs, and a pitch of 1.5, followed by PET acquisition from the mid-thigh to skull-base, 3 minutes each bed. After image acquisition, the subject will be observed for half an hour, and will be discharged if no adverse event happens.
  The estimated organ doses show that the kidneys and the urinary bladder wall were the organs with the highest dose. As presented, the effective doses for patients were 0.023 mSv/MBq ± 15% (maximum deviation), leading to an effective dose of 3.4 mSv for an injected activity of 150 MBq.
  Other Names: Ga-68 PSMA-11, PSMA-HBED-CC

SUMMARY:
This is an open-label single arm clinical trial, plan to enroll approximately a total of 62 evaluable subjects. According to the estimated missing rate 15%, the sample size in this study is 73.

Inclusion criteria:

To be eligible for inclusion, each patient must fulfill all of the following criteria:

1. Age equals or more than 20 years old
2. Willing to sign the informed consent
3. Pathology-proved intermediate to high risk group prostate cancer patients (PSA > 10 ng/mL, or Gleason score 7-10, or clinical stage >T2a) OR Prior radiotherapy or prostatectomy for prostate cancer with biochemical recurrence defined as:

   * post prostatectomy: increase in PSA of > 0.2 ng/mL in two or more consecutive blood samples
   * post radiotherapy: PSA levels of ≥ 2 ng/mL above the post-therapy nadir
4. Life expectancy more than 3 months

Exclusion criteria:

Patient who has any of the following criteria will be excluded from the trial:

1. Unable to tolerate the PET/CT scan, such as those with claustrophobia, unable to lie still, consciousness unclear, vital sign unstable.
2. With renal impairment (glomerular filtration rate lower than 30 ml/min/1.73 m2), and allergy to medium contrast
3. Unable to give informed consent.
4. Allergy history to Ga68-PSMA ligand, significant abnormal lab data (ALT more than three times of normal value), and high risk to conduct examination after evaluations of PI.
5. Patient had malignancy history

DETAILED DESCRIPTION:
It is a phase II single-arm clinical trial. The primary endpoint is diagnostic sensitivity of the Ga-68 PSMA ligand in prostate cancer. The four outcomes (true positive, false positive, true negative, and false negative) can be defined based on the process as Figure 1 and formulated in a 2×2 contingency table, and the related sensitivity, specificity, and accuracy will be calculated based on the test results of enrolled subjects. All subjects enrolled must meet eligibility criteria based on the inclusion/exclusion criteria detailed in Section 5.4 and 5.5.

Time elapsed from the last PSA determination until PET was no more than 2 weeks in all patients. Patients will receive complementary workups including MRI (for patients suspicious for local or regional node recurrence), bone scan (for patients suspicious for distant bone metastasis), contrast CT (for patients suspicious for visceral organ metastasis or lung metastasis) subsequently after Ga68-PSMA ligand PET/CT scan no longer than two weeks.

All of the images were interpreted by a team of two nuclear medicine physicians and one radiologist. In cases of questionable findings, the decision was made by consensus of at least two observers using pre-specified criteria. All of the readers were blinded to the patient's clinical history, blood tests, and previous imaging findings. If patient have consistent findings between Ga68 PSMA ligand PET/CT and other complementary workups, the patients are deemed as true positive or negative. For patients with discrepancy image findings between Ga68 PSMA ligand PET/CT and the other complementary workups, biopsy, needle aspiration or operation will be arranged for histology confirmation. The final results of Ga68-PSMA ligand PET/CT scan will be depend on the consensus of multidisciplinary tumor board based on all integrated informations.

ELIGIBILITY:
Inclusion Criteria:

1. Age equals or more than 20 years old
2. Willing to sign the informed consent
3. Pathology-proved intermediate to high risk group prostate cancer patients (PSA > 10 ng/mL, or Gleason score 7-10, or clinical stage >T2a) OR Prior radiotherapy or prostatectomy for prostate cancer with biochemical recurrence defined as:

   * post prostatectomy: increase in PSA of > 0.2 ng/mL in two or more consecutive blood samples
   * post radiotherapy: PSA levels of ≥ 2 ng/mL above the post-therapy nadir

Exclusion Criteria:

1. Unable to tolerate the PET/CT scan, such as those with claustrophobia, unable to lie still.
2. With renal impairment (glomerular filtration rate lower than 30 ml/min/1.73 m2), and allergy to medium contrast
3. Unable to give informed consent.
4. Allergy history to Ga68-PSMA ligand, significant abnormal lab data, and high risk to conduct examination after evaluations of PI.

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Ga-68 PSMA ligand : A radiopharmaceutical for localization of prostate cancer | Three years
  To evaluate sensitivity of Ga68 PSMA ligand compared with a reference value of the standard

CONTACTS AND LOCATIONS:
Overall Officials: Tseng Jing-Ren, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital ,Linkou, Taoyuan, Taiwan